CLINICAL TRIAL: NCT01583244
Title: Korean Post-marketing Surveillance for Orencia®
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-300
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with active rheumatoid arthritis: Patients aged 6 years and over who have moderate-to-severe active rheumatoid arthritis
  Interventions: Drug: No Intervention (subjects were previously treated with Orencia®)

INTERVENTIONS:
Drug: No Intervention (subjects were previously treated with Orencia®) — No Intervention
  Other Names: Abatacept

SUMMARY:
The purpose of this post-marketing surveillance is to investigate and confirm the type and incidence of newly identified adverse events and any other factors affecting safety and efficacy of Orencia® so that the regulatory authority can manage the marketing approval properly.

DETAILED DESCRIPTION:
Time Perspective: Prospective / Retrospective(On-treatment)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients must be diagnosed with: Adult Rheumatoid arthritis (RA): adult patients with moderate-to-severe active RA

Or

* Juvenile idiopathic RA: juvenile patients aged 6 years and older with moderate-to-severe active RA

Exclusion Criteria:

* Children aged <6 years
* Pregnant or lactating women
* Patients who are participating in another study
* Patients known to be hypersensitive to the active component of the surveillance drug or any other component of the surveillance drug
* Patients who had a positive tuberculosis screening test but were not treated with standard therapy before participating in the study
* Patients who have a positive hepatitis virus test
* Patients who were given a live vaccine concurrently with the surveillance drug or are expected to be given a live vaccine again within 3 months after discontinuation of the surveillance drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 6 years and over who have moderate-to-severe active rheumatoid arthritis
Sampling Method: Non-Probability Sample
Enrollment: 701 (Actual)
Dates: Start 2010-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Adverse events occurrence | 30 days after last dose of study drug

SECONDARY OUTCOMES:
Number of Adverse Events and Serious Adverse Events | 30 days after last dose of study drug
Efficacy of Orencia® measured by swollen joint counts and tender joint counts in the subject treated with the surveillance drug, patient-assessed pain, APR, patient-assessed global health, physician-assessed global disease activity | 24 weeks of registration
  * APR = acute phase reactants

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Seoul, South Korea

REFERENCES:
- [Derived] Lee JS, Ahmad H, Shim SC, Bae SC, Song YW, Lee EY. High Proportion of Subjective Component to the Disease Activity Score is Associated with Favorable Response to Abatacept in Rheumatoid Arthritis. Patient. 2019 Jun;12(3):319-326. doi: 10.1007/s40271-018-0347-z. PMID 30484084
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx